CLINICAL TRIAL: NCT00255073
Title: Does Reducing Spasticity Permit an Increase in Strength?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Terence Sanger, Associate Professor, University of Southern California
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BACLOFEN
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Spastic Diplegic Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Baclofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: baclofen

SUMMARY:
Reduction of spasticity has been a major focus of the treatment of childhood cerebral palsy, resulting in numerous treatment strategies that target various parts of the motor system. However, in many children weakness may be a greater contributor to disability than spasticity. Recent results suggest a correlation between spasticity and weakness, but it is not known if reduction of spasticity can improve strength.

We suggest a simplified model in which spinal mechanisms (including reflex contributions to spasticity) and supraspinal mechanisms (including voluntary contributions to strength) combine to activate muscle. The model implies that the supraspinal contribution cannot increase unless the spinal contribution decreases. We therefore hypothesize that reduction of spasticity improves the ability to increase voluntary strength.

We propose a double-masked placebo-controlled clinical trial combining treatment using the oral anti-spasticity medication baclofen with a 6-week program of strength training. We will enroll 20 ambulatory children with spastic diplegic cerebral palsy. Prior to and following the intervention, we will obtain quantitative measures of spasticity, strength, and gait. We predict that the children taking baclofen will have a greater increase in strength than the children taking placebo. We predict that the increase in strength will be reflected in improved performance on gait analysis, and it will correlate with a reduction in quantitative measures of spasticity and spinal reflex excitability.

If the hypothesis is correct, it will provide important new information on the relationship between spasticity and strength in children with cerebral palsy. It will provide the first measurements of the effect of baclofen on voluntary muscle activation in children. It will support the short-term use of combined anti-spasticity medication and strengthening as a new clinical treatment for ankle weakness in children with spastic diplegia. A successful result will have immediate and significant implications for treatment of children with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosis of Cerebral Palsy 2. Spasticity at extensor muscle groups of one or both ankles according to the definition of the Task Force on Childhood Motor Disorders, and as evidenced by the presence of a spastic catch or velocity-dependent hypertonia on rapid passive muscle lengthening while the subject attempts to maintain a relaxed state 3. Ambulatory without assistive devices 4. Sufficient ability to follow instructions to be able to comply with the strengthening program and strength testing

Exclusion Criteria:

* 1. Contracture at the ankle, or a limitation of the passive range of motion such that neutral position is not achievable with the knee extended.

  2. Hypersensitivity or allergy to Baclofen or related medications, or any medical condition that would be expected to increase the risks of this study 3. Respiratory difficulty due to weakness, restrictive lung disease, obstructive lung disease, tracheomalacia, or laryngeal weakness 4. Renal failure or chronic kidney disease 5. Pregnancy or planned pregnancy (sexually active girls will be asked to take a urine pregnancy test prior to study entry) 6. Difficulty maintaining head position while standing or seated 7. Current use of other anti-spasticity agents, including valium, tizanidine, clonidine, dantrolene, or similar agents 8. Use of oral baclofen within 3 months prior to study entry 9. Injection of botulinum toxin into the calf muscles within 3 months prior to study entry 10. Prior implantation of a baclofen pump or deep-brain stimulator 11. Seizure within previous two years 12. Lower extremity dystonia 13. Bradykinesia or evidence of parkinsonism 14. Spinal cord injury 15. Neurodegenerative disease 16. Ankle, foot, lower leg, or Achilles tendon surgery within the previous year 17. Dorsal rhizotomy or neurotomy

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10
Dates: Start 2005-01; Study Completion 2006-04

PRIMARY OUTCOMES:
Maximal Voluntary Contraction

SECONDARY OUTCOMES:
H reflex

CONTACTS AND LOCATIONS:
Overall Officials: Terence Sanger, md,phd, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States